CLINICAL TRIAL: NCT00232648
Title: Investigation of Safety and Efficacy of Budesonide Inhalation Suspension in the Long-Term Use in Japanese Children With Bronchial Asthma (Open Long-Term Extension Study Following Study SD-004-0765
Brief Title: Long Term Safety & Efficacy of Budesonide Inhalation Suspension in Japanese Children With Bronchial Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SD-004-0768
Record Dates: First submitted 2005-09-30; First posted 2005-10-05 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide

INTERVENTIONS:
Drug: Pulmicort (budesonide) Respules

SUMMARY:
This study is as an extension study of SD-004-0765, to assess the safety profile of long-term use of budesonide inhalation suspension in Japanese young children with bronchial asthma. Children completing study SD-004-0765 continued administration of budesonide inhalation suspension as judged by the investigator; the dose is adjusted as appropriate within the range of 0.25 to 1.0 mg per day administered once or twice daily, according to the symptoms.

ELIGIBILITY:
Inclusion Criteria:

- 1. Clinical benefit from continued treatment with budesonide inhalation suspension was expected in patients with bronchial asthma participating in study SD-004-0765, as judged by the investigator(s) at the completion of that study (Visit 11, Week 24), and the patient's caregiver wished the continued treatment with budesonide inhalation suspension A written consent to participate in this study had been obtained from the patient's legal representative (a person who exercises parental authority for the patient, or if no one was applicable, a guardian: in principle, the patient's parent).

3. The patient was younger than 5 years old. Patients aged 5 years could be included in this study if no other effective treatment for the patient's bronchial asthma was available as judged by the investigator(s).

Exclusion Criteria:

-1. Concurrent severe diseases of liver, kidney, heart or other complications. 2. Contra-indications (eg, known or suspected allergy) to budesonide or excipients contained in the investigational product.

3. Other conditions, in which the investigator(s) judges patient's participation in this study inappropriate.

Ages: 13 Months to 65 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54
Dates: Start 2004-01; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
The safety profile of long-term use of budesonide inhalation suspension assessed by evaluation of frequency and intensity of adverse events, plasma cortisol, physical examination, height, weight and clinical laboratory values.

SECONDARY OUTCOMES:
The efficacy of budesonide inhalation suspension assessed by overall evaluation on asthma control by investigator

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca KK RITA Medical Director, Study Director — AstraZeneca KK - Pharmaceuticals
Locations (9):
- Japan (9):
  - Fukuoka, Fukuoka
  - Isehara, Kanagawa
  - Tsu, Mie-ken
  - Kurashiki, Okayama-ken
  - Hioshima
  - Kanagawa
  - Matsuyama
  - Obhu-city
  - Tokyo